CLINICAL TRIAL: NCT00970710
Title: Vaasa Childhood Obesity Primary Prevention Study
Acronym: VACOPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Foundation for Paediatric Research, Finland (Other); Vaasa Health care center (Unknown); Seinajoki Central Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Taina Mustila, M.D. Ph.D., Seinajoki Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 100454
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Childhood Obesity Pevention

STUDY DESIGN:
Intervention Model Description: Pragmatic controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle counseling (Experimental): VACOPP (Vaasa Childhood Obesity Primary Prevention Study): Intensified lifestyle counseling including physical activity and nutritional information beginning during maternity health care and continuing during child health care clinic visits.
  Interventions: Behavioral: Vaasa Childhood Obesity Primary Prevention Study

INTERVENTIONS:
Behavioral: Vaasa Childhood Obesity Primary Prevention Study — Intensified counselling concerning healthy diet and suitable physical activity during pregnancy to mothers in the intervention group continuing in child health care clinic visits with the offspring until child's age of 5 year.
  Other Names: VACOPP

SUMMARY:
This study aims to prevent childhood obesity with early life (pregnancy) intensified counselling. The recruited intervention group is pregnant mothers who are at risk to get gestational diabetes. Lifestyle intervention (nutritional and physical activity) begins during pregnancy in maternity clinics and continues in child wellfare clinics until the child is 5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are at risk to get gestational diabetes.

Exclusion Criteria:

* Foreigner with language problems
* Major psychosocial problems
* Diabetes mellitus type I or II
* Physical disability,
* Major medical problems in pregnancy

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Preventing childhood obesity | Offspring age until six years
  Difference in offspring weight gain compared to control group

SECONDARY OUTCOMES:
lower cholesterol values | up to six years
lower HOMA-index | up to six years

CONTACTS AND LOCATIONS:
Overall Officials: Taina E. Mustila, M.D. Ph.D., Principal Investigator — Seinajoki Central Hospital
Locations (1):
- Health care center in Vaasa, Vaasa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mustila T, Raitanen J, Keskinen P, Luoto R. A pragmatic controlled trial to prevent childhood obesity within a risk group at maternity and child health-care clinics: results up to six years of age (the VACOPP study). BMC Pediatr. 2018 Feb 27;18(1):89. doi: 10.1186/s12887-018-1065-3. PMID 29486763
- [Derived] Mustila T, Raitanen J, Keskinen P, Saari A, Luoto R. Pragmatic controlled trial to prevent childhood obesity in maternity and child health care clinics: pregnancy and infant weight outcomes (the VACOPP Study). BMC Pediatr. 2013 May 20;13:80. doi: 10.1186/1471-2431-13-80. PMID 23688259
- [Derived] Mustila T, Keskinen P, Luoto R. Behavioral counseling to prevent childhood obesity--study protocol of a pragmatic trial in maternity and child health care. BMC Pediatr. 2012 Jul 3;12:93. doi: 10.1186/1471-2431-12-93. PMID 22759439
- Available data/document: Study Protocol — http://bmcpediatr.biomedcentral.com/articles/10.1186/1471-2431-12-93
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/?term=mustila+taina+vacopp